CLINICAL TRIAL: NCT06617741
Title: Myasthenia Gravis Foundation of America Global MG Patient Registry
Acronym: MGFAPR
Status: Recruiting | Type: Observational
Sponsor: Myasthenia Gravis Foundation of America (Other)
Collaborators: Alira Health (Other)
Responsible Party: Sponsor
Other Study IDs: X130401004
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Myasthaenia Gravis; Myasthenia; Myasthenia Gravis Associated with Thymoma; Myasthenia Gravis Crisis; Myasthenia Gravis Exacerbations; Myasthenia Gravis Generalised; Myasthenia Gravis with Exacerbation (Disorder); Myasthenia Gravis, Adult Form; Myasthenia Gravis, Generalized; Myasthenia Gravis, Ocular; Myasthenia Gravis, Thymectomy; Myasthenia Gravis; Myasthenia Gravis, MuSK
Keywords: myasthenia; patient registry; MGFA; Myasthenia Gravis Foundation of America; myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants: Those with Myasthenia Gravis

SUMMARY:
The goal of this observational study is to learn about the experiences of people living with Myasthenia Gravis (MG) in the United States. The main questions it aims to answer are:

* How and when are people with MG diagnosed?
* What are the most common symptoms associated with MG?
* What treatments are being used to treat MG?
* What are the impacts of MG on activities of daily living, employment and quality of life?
* What are the experiences with exacerbation, hospitalization and healthcare access for people with MG? Participants will answer a survey to enroll in the study, and be invited to fill out an update survey twice a year.

DETAILED DESCRIPTION:
This is a longitudinal, observational, patient reported registry.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* positive MG diagnosis

Exclusion Criteria:

* age under 18
* misdiagnosed with MG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with access to a mobile device or desktop computer with internet connection are eligible to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Estimated)
Dates: Start 2013-10-12 (Actual); Primary Completion 2029-09-19 (Estimated); Study Completion 2029-09-19 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of MG | At enrollment
  Whether the patient has a confirmed MG diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Patient Registry PI, Principal Investigator — Yale University
Locations (1):
- Myasthenia Gravis Foundation of America, Westborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Direct access to IPD is not widely shared. However, analysis of the data can be facilitated through collaboration with Alira Health.